CLINICAL TRIAL: NCT05131087
Title: A First-In-Human Clinical Trial to Evaluate the Safety, Effectiveness and Surgical Characteristics of CADENCE in Patients With Refractory Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF8-CL-20-02
Record Dates: First submitted 2021-11-02; First posted 2021-11-23 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma
Keywords: glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cadence (Experimental): Cadence procedure
  Interventions: Device: Cadence implant

INTERVENTIONS:
Device: Cadence implant — CADENCE Glaucoma Drainage Device System is a single use implantable glaucoma drainage device used for the surgical treatment of refractory glaucoma. The device is implanted in the eye using an ab-externo approach

SUMMARY:
To evaluate safety, effectiveness, and the surgical performance of CADENCE in patients with refractory glaucoma.

DETAILED DESCRIPTION:
CADENCE a single use implantable glaucoma drainage device used for the surgical treatment of refractory glaucoma. The device is implanted in the eye using an ab-externo approach

ELIGIBILITY:
Inclusion Criteria:

* 22-80 years of age.
* moderate to severe refractory glaucoma
* Able to consent

Exclusion Criteria:

* Women of child-bearing potential
* Intraocular surgery or laser within the last 3 months
* Ocular infection or inflammation within the last 6 months or currently active
* Current use of anti-coagulant therapy
* History of bleeding disorder or coagulopathies
* Subject plans to undergo any ocular surgery (including cataract surgery) during the study period
* History of corneal transplantation
* History of ICE Syndrome or epithelial ingrowth/downgrowth
* History of congenital glaucoma
* Elevated episcleral venous pressure

  -. Persistent angle closure-
* Previous glaucoma filtration surgery- -Presence of conjunctival scarring -
* neovascular glaucoma
* AC lens or scleral sutured IOL
* Aphakia
* inability to DC contact lenses
* Presence of intraocular silicone oil
* Vitreous in AC

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Assessment of AEs | 12 months
  comparison of intra-operative and post-operative adverse events observed to events reported in published literature,

SECONDARY OUTCOMES:
Surgical Experience Evaluation | 12 months
  An evaluation of the surgical experience using feedback questionnaire to describe specific note of performance characteristics of each implant.
Change in IOP | 12 months
  Change in IOP from Screening to M12
Change in IOP Lowering Medications | 12 months
  Change in IOP lowering medications from Screening to M12

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sun, PhD, Study Director — New World Medical, Inc.
Locations (1):
- Clinica Laser y Ultrasonido Ocular de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No